CLINICAL TRIAL: NCT00838747
Title: Measurement of the Folate Receptor in Blood
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR3028
Record Dates: First submitted 2008-09-05; First posted 2009-02-06 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: folate receptor; blood samples; ovarian cancer; development of measure of folate receptor in blood samples; possible selection of patients for treatment with FR targeted agents
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gynaecological Cancer: Gynaecological Cancer

SUMMARY:
The folate receptor (FR) is a cell marker that is over expressed on the cell surface of certain cancers, this occurs most frequently in ovarian cancers. Some normal tissues also express the FR, however in these normal tissues the FR is usually located on the tissue surface that is inaccessible to circulating drugs. As such, drugs which target the FR may potentially be used to achieve anti-tumour efficacy whilst reducing toxicity to normal tissues. Therefore the ability to measure FR levels from different cancer types may help to select patients who are most likely to benefit from treatment with FR targeted therapies. One such drug BGC 945 is currently being tested in preclinical study at The Institute of Cancer Research

DETAILED DESCRIPTION:
A method has been developed in the laboratory which has been able to measure FR obtained from cancer cells in culture that has been added into blood. We would like to study if this method can measure FR in plasma and serum obtained from patients with ovarian cancer. We would also like to analyse plasma and serum samples obtained from healthy volunteers to determine if they have any appreciable levels of FR, which can then be compared to the measurements obtained from cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage III/IV ovarian cancer
* healthy volunteers who are staff at the ICR and RMH

Exclusion Criteria:

* patients or healthy volunteers who are unable to give informed consent
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To measure the levels of folate receptor in blood samples obtained from patients with ovarian cancer and from healthy volunteers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stan Kaye, Professor, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, Sutton, United Kingdom